CLINICAL TRIAL: NCT05150340
Title: A Phase 3, Open-label, Non-controlled Study to Evaluate the Pharmacokinetics, Safety and Tolerability, and Efficacy of TAK-771 in Japanese Subjects With Primary Immunodeficiency Diseases (PID)
Brief Title: A Study of TAK-771 in Japanese People With Primary Immunodeficiency Diseases (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-771-3004; jRCT2031210457 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epoch 1: TAK-771 Ramp up Period (Experimental): TAK-771 included IGI 10% and Recombinant Human Hyaluronidase (rHuPH20). Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution. The dose of 10% IGI was increased from 1/3 of full dose to full dose in 3 weeks for participants who received TAK-771 once every 3 weeks, or from 1/4 of full dose to full dose in 6 weeks for participants who received TAK-771 once every 4 weeks.
  Interventions: Drug: TAK-771
- Epoch 2: TAK-771 Full Dose Treatment Period (Experimental): TAK-771 included Immune Globulin Infusion (IGI) 10% and Recombinant Human Hyaluronidase (rHuPH20). Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3, or 4 weeks for up to Week 27 for participants with 4-Week dosing interval or Week 25 for participants with 3-Week dosing interval.
  Interventions: Drug: TAK-771

INTERVENTIONS:
Drug: TAK-771 — Intervention description; Immune Globulin Infusion (IGI) 10% and Recombinant Human Hyaluronidase (rHuPH20)
  Other Names: Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase

SUMMARY:
The main aim of the study is to check how much TAK-771 stays in their blood over time, side effect from the study treatment or TAK-771, how much TAK-771 participants can receive without getting side effects from it, and if TAK-771 improves symptoms of primary immunodeficiency diseases (PID). This will help the study sponsor (Takeda) to work out the best dose to give people in the future.

The participants will be treated with TAK-771 for totally 27 or 30 weeks. Treatment period is consist of two periods called Epoch 1 and Epoch 2. In Epoch 1, different groups of participants will receive lower to higher doses of TAK-771 for 3 to 6 weeks. The study doctors will check for side effects from each dose of TAK-771. In Epoch 2, participants will receive TAK-771 once a 3 or 4 weeks until the end of 24 weeks.

There will be many clinic visits. The number of visits will depend on the infusion cycles of study drug (every 3, or 4 weeks).

ELIGIBILITY:
Inclusion Criteria

1. Be a Japanese person.
2. Participant must have a documented diagnosis of a form of primary humoral immunodeficiency involving antibody formation and requiring gammaglobulin replacement, as defined according to the International Union of Immunological Societies(IUIS) Committee 2017. The diagnosis must be confirmed by the Medical Director prior to TAK-771 treatment.
3. Participant has been receiving a stable clinical dose of intravenous immunoglobulin (IVIG) or conventional subcutaneous immunoglobulin (cSCIG), which is equivalent to approximately 200 to 600 mg/kg body weight per 3 to 4 week period for IVIG and approximately 50 to 200 mg/kg body weight per week for cSCIG based on the description in the package insert, consistently over a period of at least 3 months prior to screening, or Participant has been receiving of TAK-664 with fixed dose and dosing frequency at least 3 months prior to enrollment. That is, participant is about to complete Study TAK-664-3001 or participating in Study TAK-664-3002.
4. Participant who has been receiving IVIG or cSCIG had all serum trough levels of total immunoglobulin G (IgG) >=5 g/L within 1 month prior to the screening/enrollment.
5. Serum trough levels at screening/enrollment meet one of the following:

   1. IVIG-treated or cSCIG-treated participants Participant who had serum trough levels of IgG >=5 g/L at the last 2 points in screening procedure before the first administration of TAK-771.
   2. TAK-664-treated participants Participant who had serum trough levels of IgG >=5 g/L at the last 2 points in TAK-664 studies before the first administration of TAK-771.
6. Participant is willing and able to comply with use of digital tools and applications.

Exclusion Criteria

1. Participant has a known history of or is positive at screening/enrollment for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2 For participants who are switching from TAK-664 studies, the eligibility will be reconfirmed after result of the specialty test conducted at Week 1 become available.
2. Abnormal laboratory values at screening/enrollment meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

   * Persistent alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 times the upper limit of normal (ULN) for the testing laboratory
   * Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] =<500/mm^3)
3. Participant has presence of renal function impairment defined by eGFR <60 mL/min/1.73m^2.
4. Participant has been diagnosed with, or had a malignancy (other than adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the disease-free period prior to screening exceeds 5 years.
5. Participant is receiving anti-coagulation therapy or has a history of thrombotic episodes (including deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism) within 12 months prior to screening/enrollment or a history of thrombophilia.
6. Participant has abnormal protein loss (protein losing enteropathy, nephrotic syndrome)
7. Participant has anemia that would preclude phlebotomy for laboratory studies according to standard practice at the site.
8. Participant has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IVIG, subcutaneous immunoglobulin (SCIG), and/or Immune Serum Globulin infusions
9. Participant has immunoglobulin A (IgA) deficiency (serum IgA less than 0.07g/L) and history of hypersensitivity, or history of confirmed anti-IgA antibodies, or both.
10. Participant is on preventative (prophylactic) systemic antibacterial antibiotics at doses sufficient to treat or prevent bacterial infections, and cannot stop these antibiotics at the time of screening/enrollment.
11. Participant has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening/enrollment or had a serious bacterial infection within the 3 months prior to screening/enrollment
12. Participant has a bleeding disorder, or a platelet count less than 20,000/microL, or in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of subcutaneous (SC) therapy.
13. Participant has total protein >9 g/dL or myeloma, or macroglobulinemia (IgM) or paraproteinemia.
14. Participant has a known allergy to hyaluronidase
15. Participant has severe dermatitis that would preclude adequate sites for safe product administration.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- Japan (12):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hospital of University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Shinshu University Hospital, Matsumoto, Nagano
  - Tokyo Medical Dental University Hospital, Bunkyo-ku, Tokyo
  - National Center for Child Health and development, Setagaya-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima University Hospital, Hiroshima
  - Saitama Prefectual Children's Medical Center, Saitama
  - Shizuoka Childrens Hospital, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/61b2391cf571d4002a64b47b

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a confirmed diagnosis of primary immunodeficiency diseases (PID) took part in the study at 12 investigative sites in Japan from 24 January 2022 to 28 August 2023.
Pre-assignment Details: Participants with PID, who had been receiving a consistent dose of intravenous immunoglobulin (IVIG), conventional subcutaneous immunoglobulin (cSCIG) or TAK-664 (immune globulin subcutaneous [human], 20% solution [20%SCIG]) for at least 3 months prior to screening were enrolled in the study to receive TAK-771.
Period: Epoch 1
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Started | 16 | 0
Pharmacokinetic Analysis Set 1 (Pharmacokinetic Analysis Set 1 included participants for analysis of total serum IgG trough levels for total serum levels of IgG and IgG subclasses.) | 16 | 0
Pharmacokinetic Analysis Set 2 (Pharmacokinetic analysis set 2 included the analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2 participants. (N=16). There were 4 participants aged 12 years or older who consented to blood sampling for analysis of PK parameters, and Pharmacokinetic Analysis Set 2 analysis was performed on a subset consisting of these 4 participants.) | 0 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Epoch 2
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Started | 0 | 16
Pharmacokinetic Analysis Set 1 (Pharmacokinetic Analysis (PK) Set 1 included participants for analysis of total serum IgG trough levels for total serum levels of IgG and IgG subclasses.) | 0 | 16
Pharmacokinetic Analysis Set 2 (Pharmacokinetic analysis set 2 included the analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2 participants. (N=16). There were 4 participants aged 12 years or older who consented to blood sampling for analysis of PK parameters, and Pharmacokinetic Analysis Set 2 analysis was performed on a subset consisting of these 4 participants.) | 0 | 4
Completed | 0 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all enrolled subjects who received investigational drug at least once. Analyses of safety, tolerability and product administration were based on the SAS.
Groups:
- Epoch 1: TAK-771: TAK-771 included IGI 10% and rHuPH20. Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution. The dose of 10% IGI was increased from 1/3 of full dose to full dose in 3 weeks for participants who received TAK-771 once every 3 weeks, or from 1/4 of full dose to full dose in 6 weeks for participants who received TAK-771 once every 4 weeks.
Arm/Group | Epoch 1: TAK-771
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.2 (16.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 16
Height at Baseline [Mean (Standard Deviation); unit: Centimeters (cm)] | 149.26 (25.892)
Weight at Baseline [Mean (Standard Deviation); unit: Kilograms (kg)] | 44.33 (16.509)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI=weight (kg) / [height (m)]^2
  kilograms per meter square (kg/m^2) | 19.05 (2.747)

OUTCOME MEASURES:

1. Primary Outcome: Epoch 2: Serum Trough Levels of Total IgG Antibodies After Administration of TAK-771
Description: The data was reported at Week 7, 11, 15, 19, 23, 27, and 31 for 4-Week interval and at Week 4, 7, 10, 13, 16, 19, 22, 25 and 28 for 3-Week interval.
Time Frame: Up to Week 31 for Participants with 4-Week Dosing Interval or Up to Week 28 for Participants with 3-Week Dosing Interval
Population: PK analysis set: all enrolled participants who received investigational drug once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect serum IgG concentration analysis results. PK set 1: analysis of total serum IgG trough levels for total serum levels of IgG and IgG subclasses. Overall number analyzed: number of participants available for analysis. Number analyzed: participants with data available for analysis at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams/Liter (g/L)
Groups:
- Epoch 2: TAK-771 Full Dose Treatment Period: TAK-771 included IGI 10% and rHuPH20. Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3, or 4 weeks for up to Week 27 for participants with 4-Week dosing interval or Week 25 for participants with 3-Week dosing interval.
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
grams/Liter (g/L)
  Week 7, 4-Week Interval: number analyzed (Participants) | 12
  Week 7, 4-Week Interval | 9.372 (10.3)
  Week 11, 4-Week Interval: number analyzed (Participants) | 12
  Week 11, 4-Week Interval | 8.741 (13.7)
  Week 15, 4-Week Interval: number analyzed (Participants) | 11
  Week 15, 4-Week Interval | 8.929 (13.0)
  Week 19, 4-Week Interval: number analyzed (Participants) | 12
  Week 19, 4-Week Interval | 9.150 (15.5)
  Week 23, 4-Week Interval: number analyzed (Participants) | 12
  Week 23, 4-Week Interval | 8.944 (20.9)
  Week 27, 4-Week Interval: number analyzed (Participants) | 11
  Week 27, 4-Week Interval | 9.006 (18.4)
  Week 31, 4-Week Interval: number analyzed (Participants) | 12
  Week 31, 4-Week Interval | 9.159 (20.8)
  Week 4, 3-Week Interval: number analyzed (Participants) | 2
  Week 4, 3-Week Interval | 13.51 (29.7)
  Week 7, 3-Week Interval: number analyzed (Participants) | 2
  Week 7, 3-Week Interval | 13.15 (35.7)
  Week 10, 3-Week Interval: number analyzed (Participants) | 2
  Week 10, 3-Week Interval | 12.54 (43.2)
  Week 13, 3-Week Interval: number analyzed (Participants) | 0
  Week 16, 3-Week Interval: number analyzed (Participants) | 2
  Week 16, 3-Week Interval | 13.50 (39.7)
  Week 19, 3-Week Interval: number analyzed (Participants) | 2
  Week 19, 3-Week Interval | 12.76 (46.9)
  Week 22, 3-Week Interval: number analyzed (Participants) | 2
  Week 22, 3-Week Interval | 12.79 (40.1)
  Week 25, 3-Week Interval: number analyzed (Participants) | 2
  Week 25, 3-Week Interval | 12.95 (57.6)
  Week 28, 3-Week Interval: number analyzed (Participants) | 2
  Week 28, 3-Week Interval | 12.70 (43.0)

2. Secondary Outcome: Epoch 2: Maximum Concentration (Cmax) of Total Serum Levels of IgG and IgG Subclasses
Time Frame: Pre-infusion at Week 27 for participants with 4-Week or Week 25 with 3-Week dosing interval and post infusion at multiple time points up to Week 31 for participants with 4-Week dosing interval and up to Week 28 with 3-Week dosing interval.
Population: Pharmacokinetic analysis set included all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. Pharmacokinetic analysis set 2 included the analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/L
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
g/L
  Total IgG | 12.72 (23.4)
  IgG Subclass (IgG 1) | 7.694 (16.7)
  IgG Subclass (IgG 2) | 4.140 (23.0)
  IgG Subclass (IgG 3) | 0.2396 (46.7)
  IgG Subclass (IgG 4) | 0.3200 (36.3)

3. Secondary Outcome: Epoch 2: Time to Maximum Concentration (Tmax) of Total Serum Levels of IgG and IgG Subclasses (IgG1, IgG2, IgG3, and IgG4)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
days
  Total IgG | 6.94 [2.94 to 8.85]
  IgG Subclass (IgG 1) | 3.92 [2.94 to 8.83]
  IgG Subclass (IgG 2) | 3.92 [2.94 to 8.83]
  IgG Subclass (IgG 3) | 2.99 [2.80 to 8.83]
  IgG Subclass (IgG 4) | 3.88 [2.80 to 5.04]

4. Secondary Outcome: Epoch 2: Area Under the Curve (AUC) of Total Serum Levels of IgG and IgG Subclasses (IgG1, IgG2, IgG3, and IgG4)
Description: AUC is expressed as grams*day per liter/grams per kilograms [(g*day/L)/(g/kg)].
Time Frame: as for outcome 2
Population: PK analysis set: all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK analysis set 2: analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2. Number of participants analyzed are number of participants available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (g*day/L)/(g/kg)
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
(g*day/L)/(g/kg)
  Total IgG, AUCtau/Dose: number analyzed (Participants) | 3
  Total IgG, AUCtau/Dose | 767.9 (40.0)
  Total IgG, AUClast/Dose | 625.6 (55.2)
  IgG Subclass (IgG 1), AUCtau/Dose | 432.4 (36.2)
  IgG Subclass (IgG 1), AUClast/Dose | 370.7 (53.0)
  IgG Subclass (IgG 2), AUCtau/Dose | 230.4 (25.2)
  IgG Subclass (IgG 2), AUClast/Dose | 197.4 (40.5)
  IgG Subclass (IgG 3), AUCtau/Dose | 7.916 (165.6)
  IgG Subclass (IgG 3), AUClast/Dose | 5.449 (227.2)
  IgG Subclass (IgG 4), AUCtau/Dose | 15.65 (37.1)
  IgG Subclass (IgG 4), AUClast/Dose | 12.08 (53.4)

5. Secondary Outcome: Epoch 2: Half-life of Total Serum Levels of IgG and IgG Subclasses (IgG1, IgG2, IgG3, and IgG4)
Time Frame: At multiple time points post-infusion from Week 7 for participants with 4-Week or Week 4 with 3-Week dosing interval up to Week 31 for participants with 4-Week dosing interval and up to Week 28 with 3-Week dosing interval
Population: PK analysis set: all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK analysis set 2: analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2. Number of participants analyzed is number of participant available for analysis.
Measure: Median (Full Range); unit: day
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
day
  Total IgG: number analyzed (Participants) | 1
  Total IgG | NA [NA to NA] — Data was not calculated due to <3 contributes based on the analysis plan for this outcome measure.
  IgG Subclass (IgG 1): number analyzed (Participants) | 3
  IgG Subclass (IgG 1) | 59.7 [40.4 to 77.9]
  IgG Subclass (IgG 2): number analyzed (Participants) | 3
  IgG Subclass (IgG 2) | 49.6 [40.8 to 71.4]
  IgG Subclass (IgG 3): number analyzed (Participants) | 2
  IgG Subclass (IgG 3) | NA [NA to NA] — Data was not calculated due to <3 contributes based on the analysis plan for this outcome measure.
  IgG Subclass (IgG 4): number analyzed (Participants) | 3
  IgG Subclass (IgG 4) | 35.9 [35.8 to 46.3]

6. Secondary Outcome: Epoch 2: Apparent Total Clearance (CL/F) of Total Serum Levels of IgG and IgG Subclasses (IgG1, IgG2, IgG3, and IgG4)
Time Frame: as for outcome 2
Population: PK analysis set: all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK analysis set 2: the analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2. Number of participants analyzed is number of participants available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per day (mL/day)
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
milliliters per day (mL/day)
  Total IgG: number analyzed (Participants) | 3
  Total IgG | 76.84 (29.4)
  IgG Subclass (IgG 1) | 117.0 (37.9)
  IgG Subclass (IgG 2) | 219.6 (36.8)
  IgG Subclass (IgG 3) | 6392 (176.6)
  IgG Subclass (IgG 4) | 3234 (58.0)

7. Secondary Outcome: Epoch 2: Apparent Volume of Distribution (Vz/F) of Total Serum Levels of IgG and IgG Subclasses (IgG1, IgG2, IgG3, and IgG4)
Time Frame: as for outcome 2
Population: PK analysis set included all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK analysis set 2=analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2. Number participants analyzed: number of participants available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
mL
  Total IgG: number analyzed (Participants) | 1
  Total IgG | NA (NA) — Data was not estimable as the concentrations for all participants were below the limit of quantitation.
  IgG Subclass (IgG 1): number analyzed (Participants) | 3
  IgG Subclass (IgG 1) | 8193 (54.9)
  IgG Subclass (IgG 2): number analyzed (Participants) | 3
  IgG Subclass (IgG 2) | 14650 (57.0)
  IgG Subclass (IgG 3): number analyzed (Participants) | 2
  IgG Subclass (IgG 3) | NA (NA) — Data was not estimable as the concentrations for all participants were below the limit of quantitation.
  IgG Subclass (IgG 4): number analyzed (Participants) | 3
  IgG Subclass (IgG 4) | 165900 (88.3)

8. Secondary Outcome: Epoch 2: Minimum Concentration (Cmin) of Total Serum Levels of IgG and IgG Subclasses (IgG1, IgG2, IgG3, and IgG4)
Time Frame: as for outcome 2
Population: PK analysis set: all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect serum IgG concentration analysis results. PK analysis set 2: analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2. Number of participants analyzed: number of participants available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/L
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 4
g/L
  Total IgG | 9.347 (17.9)
  IgG Subclass (IgG 1) | 5.479 (10.7)
  IgG Subclass (IgG 2) | 2.941 (19.8)
  IgG Subclass (IgG 3): number analyzed (Participants) | 1
  IgG Subclass (IgG 3) | NA (NA) — Data was not estimable as the concentrations for participant were below the limit of quantitation.
  IgG Subclass (IgG 4): number analyzed (Participants) | 3
  IgG Subclass (IgG 4) | 0.2255 (8.4)

9. Secondary Outcome: Epoch 2: Serum Trough Levels of IgG Subclasses (IgG1, IgG2, IgG3, and IgG4) After Administration of TAK-771
Time Frame: 4-Week dosing interval (Week 7, Week 11, Week 15, Week 19, Week 23, Week 27, and Week 31); 3-Week dosing interval (Week 4, week 7, Week 10, Week 16, Week 19, Week 22, Week 25, and Week 28)
Population: PK analysis set: all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK analysis set 2: analysis of PK parameters for total serum levels of IgG, for baseline-corrected total serum levels of IgG, and for IgG subclasses in Epoch 2. Number analyzed: participants with data available for analysis at given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/L
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
g/L
  IgG 1, Week 7, 4-Week Interval: number analyzed (Participants) | 12
  IgG 1, Week 7, 4-Week Interval | 5.478 (12.1)
  IgG 1, Week 11, 4-Week Interval: number analyzed (Participants) | 12
  IgG 1, Week 11, 4-Week Interval | 5.106 (15.6)
  IgG 1, Week 15, 4-Week Interval: number analyzed (Participants) | 11
  IgG 1, Week 15, 4-Week Interval | 4.987 (11.9)
  IgG 1, Week 19, 4-Week Interval: number analyzed (Participants) | 11
  IgG 1, Week 19, 4-Week Interval | 5.063 (10.1)
  IgG 1, Week 23, 4-Week Interval: number analyzed (Participants) | 11
  IgG 1, Week 23, 4-Week Interval | 4.873 (10.8)
  IgG 1, Week 27, 4-Week Interval: number analyzed (Participants) | 11
  IgG 1, Week 27, 4-Week Interval | 5.066 (16.6)
  IgG 1, Week 31, 4-Week Interval: number analyzed (Participants) | 11
  IgG 1, Week 31, 4-Week Interval | 5.104 (14.0)
  IgG 2, Week 7, 4-Week Interval: number analyzed (Participants) | 12
  IgG 2, Week 7, 4-Week Interval | 3.147 (20.1)
  IgG 2, Week 11, 4-Week Interval: number analyzed (Participants) | 12
  IgG 2, Week 11, 4-Week Interval | 2.931 (15.0)
  IgG 2, Week 15, 4-Week Interval: number analyzed (Participants) | 11
  IgG 2, Week 15, 4-Week Interval | 2.912 (13.5)
  IgG 2, Week 19, 4-Week Interval: number analyzed (Participants) | 11
  IgG 2, Week 19, 4-Week Interval | 3.043 (16.5)
  IgG 2, Week 23, 4-Week Interval: number analyzed (Participants) | 11
  IgG 2, Week 23, 4-Week Interval | 2.976 (16.7)
  IgG 2, Week 27, 4-Week Interval: number analyzed (Participants) | 11
  IgG 2, Week 27, 4-Week Interval | 3.078 (15.5)
  IgG 2, Week 31, 4-Week Interval: number analyzed (Participants) | 11
  IgG 2, Week 31, 4-Week Interval | 3.091 (18.3)
  IgG 3, Week 7, 4-Week Interval: number analyzed (Participants) | 1
  IgG 3, Week 7, 4-Week Interval | 0.1380 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 3, Week 11, 4-Week Interval: number analyzed (Participants) | 1
  IgG 3, Week 11, 4-Week Interval | 0.1780 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 3, Week 15, 4-Week Interval: number analyzed (Participants) | 1
  IgG 3, Week 15, 4-Week Interval | 0.1390 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 3, Week 19, 4-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 23, 4-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 27, 4-Week Interval: number analyzed (Participants) | 1
  IgG 3, Week 27, 4-Week Interval | 0.2280 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 3, Week 31, 4-Week Interval: number analyzed (Participants) | 0
  IgG 4, Week 7, 4-Week Interval: number analyzed (Participants) | 12
  IgG 4, Week 7, 4-Week Interval | 0.1933 (15.9)
  IgG 4, Week 11, 4-Week Interval: number analyzed (Participants) | 12
  IgG 4, Week 11, 4-Week Interval | 0.1965 (22.7)
  IgG 4, Week 15, 4-Week Interval: number analyzed (Participants) | 11
  IgG 4, Week 15, 4-Week Interval | 0.2020 (16.8)
  IgG 4, Week 19, 4-Week Interval: number analyzed (Participants) | 11
  IgG 4, Week 19, 4-Week Interval | 0.2057 (16.1)
  IgG 4, Week 23, 4-Week Interval: number analyzed (Participants) | 11
  IgG 4, Week 23, 4-Week Interval | 0.2054 (14.6)
  IgG 4, Week 27, 4-Week Interval: number analyzed (Participants) | 11
  IgG 4, Week 27, 4-Week Interval | 0.2228 (24.6)
  IgG 4, Week 31, 4-Week Interval: number analyzed (Participants) | 11
  IgG 4, Week 31, 4-Week Interval | 0.2265 (25.6)
  IgG 1, Week 4, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 4, 3-Week Interval | 9.699 (55.6)
  IgG 1, Week 7, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 7, 3-Week Interval | 8.906 (67.0)
  IgG 1, Week 10, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 10, 3-Week Interval | 8.661 (66.7)
  IgG 1, Week 13, 3-Week Interval: number analyzed (Participants) | 0
  IgG 1, Week 16, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 16, 3-Week Interval | 8.860 (68.0)
  IgG 1, Week 19, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 19, 3-Week Interval | 8.687 (68.9)
  IgG 1, Week 22, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 22, 3-Week Interval | 8.641 (64.3)
  IgG 1, Week 25, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 25, 3-Week Interval | 8.573 (82.9)
  IgG 1, Week 28, 3-Week Interval: number analyzed (Participants) | 2
  IgG 1, Week 28, 3-Week Interval | 8.845 (68.3)
  IgG 2, Week 4, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 4, 3-Week Interval | 1.936 (105.6)
  IgG 2, Week 7, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 7, 3-Week Interval | 1.859 (89.7)
  IgG 2, Week 10, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 10, 3-Week Interval | 1.852 (83.0)
  IgG 2, Week 13, 3-Week Interval: number analyzed (Participants) | 0
  IgG 2, Week 16, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 16, 3-Week Interval | 1.964 (82.5)
  IgG 2, Week 19, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 19, 3-Week Interval | 1.944 (82.1)
  IgG 2, Week 22, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 22, 3-Week Interval | 1.957 (89.1)
  IgG 2, Week 25, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 25, 3-Week Interval | 1.910 (73.5)
  IgG 2, Week 28, 3-Week Interval: number analyzed (Participants) | 2
  IgG 2, Week 28, 3-Week Interval | 1.948 (88.1)
  IgG 3, Week 4, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 7, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 10, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 13, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 16, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 19, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 22, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 25, 3-Week Interval: number analyzed (Participants) | 0
  IgG 3, Week 28, 3-Week Interval: number analyzed (Participants) | 0
  IgG 4, Week 4, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 4, 3-Week Interval | 0.1680 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 7, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 7, 3-Week Interval | 0.1680 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 10, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 10, 3-Week Interval | 0.2010 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 13, 3-Week Interval: number analyzed (Participants) | 0
  IgG 4, Week 16, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 16, 3-Week Interval | 0.2280 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 19, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 19, 3-Week Interval | 0.2120 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 22, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 22, 3-Week Interval | 0.2230 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 25, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 25, 3-Week Interval | 0.2060 (NA) — Geometric Coefficient of variation could not be determined for single participant.
  IgG 4, Week 28, 3-Week Interval: number analyzed (Participants) | 1
  IgG 4, Week 28, 3-Week Interval | 0.2390 (NA) — Geometric Coefficient of variation could not be determined for single participant.

10. Secondary Outcome: Epoch 1 and 2: Trough Levels of Anti-Clostridium Tetani Toxoid Antibody After Administration of TAK-771
Time Frame: From Week 1, up to end of trial (EOS: Week 31 for participants with 4-Week dosing interval or Week 28 for participants with 3-Week dosing interval)
Population: PK Analysis Set included all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK Analysis Set included the analysis of total serum IgG trough levels for total serum levels of IgG and IgG subclasses. Number analyzed are number of participants with data available for analysis at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Groups:
- Epoch 1 and 2: TAK-771 included IGI 10% and Recombinant Human Hyaluronidase (rHuPH20). Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution. The dose of 10% IGI was increased from 1/3 of full dose to full dose in 3 weeks for participants who received TAK-771 once every 3 weeks, or from 1/4 of full dose to full dose in 6 weeks for participants who received TAK-771 once every 4 weeks.
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
IU/mL
  Week 1 | 1.334 (84.4)
  End of Trial (EOS): number analyzed (Participants) | 14
  End of Trial (EOS) | 1.578 (68.4)

11. Secondary Outcome: Epoch 1 and 2: Trough Levels of Anti-HBV Antibody After Administration of TAK-771
Time Frame: as for outcome 10
Population: Pharmacokinetic Analysis Set included all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect serum IgG concentration analysis results. Pharmacokinetic Analysis Set included analysis of total serum IgG trough levels for total serum levels of IgG and IgG subclasses. Number analyzed are number of participants with data available for analysis at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mIU/mL
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
mIU/mL
  Week 1 | 278.38 (125.0)
  End of Trial (EOS): number analyzed (Participants) | 14
  End of Trial (EOS) | 383.37 (57.7)

12. Secondary Outcome: Epoch 1 and 2: Trough Levels of Anti-HIB Antibody After Administration of TAK-771
Time Frame: as for outcome 10
Population: PK Analysis Set included all enrolled participants who received investigational drug at least once, have had at least 1 evaluable serum IgG concentration, and no major protocol deviations or events that would affect the serum IgG concentration analysis results. PK Analysis Set included analysis of total serum IgG trough levels for total serum levels of IgG and IgG subclasses. Number analyzed are number of participants with data available for analysis at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
ug/mL
  Week 1 | 1.958 (45.7)
  End of Trial (EOS): number analyzed (Participants) | 14
  End of Trial (EOS) | 1.519 (46.8)

13. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as Adverse events (AEs) with onset after date-time of first dose of Investigational product (IP), or medical conditions present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP.
Time Frame: From Week 1 up to Week 31 for Participants with 4-Week Dosing Interval or up to Week 28 for Participants with 3-Week Dosing Interval
Population: Safety analysis set included all enrolled participants who received investigational drug at least once. Epoch 2 Safety Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Number; unit: percentage of participants
Groups:
- Epoch 1: TAK-771 Ramp up Period: TAK-771 included IGI 10% and rHuPH20. Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution. The dose of 10% IGI was increased from 1/3 of full dose to full dose in 3 weeks for participants who received TAK-771 once every 3 weeks, or from 1/4 of full dose to full dose in 6 weeks for participants who received TAK-771 once every 4 weeks.
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants | 81.3 | 93.8

14. Secondary Outcome: Percentage of Participants With TAK-771-Related and TAK-771-Non-Related TEAEs
Description: TEAEs are defined as AEs with onset after date-time of first dose of IP, or medical conditions present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants
  TEAE Related | 56.3 | 68.8
  TEAE Non-Related | 62.5 | 81.3

15. Secondary Outcome: Percentage of Participants With Serious and Non-serious TEAEs
Description: TEAEs are defined as AEs with onset after date-time of first dose of IP, or medical conditions present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP. Serious TEAE=any untoward clinical manifestation of signs, symptoms, outcomes (related to IP or not) at any dose: results in death, was life-threatening, requires inpatient/prolongation of hospitalization, resulted in persistent/significant disability/incapacity, congenital abnormality/birth defect, important medical event. AESI=investigator-reported hypersensitivity reactions, events of disordered coagulation as bleeding/hypercoagulable AESI.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants
  Serious TEAEs | 6.3 | 6.3
  Non-serious TEAEs | 81.3 | 93.8

16. Secondary Outcome: Percentage of Participants With Severe TEAEs
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
Percentage of participants | 0 | 6.3

17. Secondary Outcome: Percentage of Participants With Local and Systemic TEAEs
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants
  Local TEAEs | 43.8 | 43.8
  Systemic TEAEs | 75.0 | 87.5

18. Secondary Outcome: Percentage of Participants With TEAEs Leading to Premature Discontinuation From Study
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants | 0 | 0

19. Secondary Outcome: Percentage of Participants With Infusion-associated TEAEs
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants | 37.5 | 50.0

20. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Clinical Laboratory Parameters Recorded as TEAEs
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants | 0 | 0

21. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Signs and Body Weight Recorded as TEAEs
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants | 0 | 0

22. Secondary Outcome: Epoch 2: Percentage of Participants Who Develop Anti-rHuPH20 Binding Antibody Titers of Greater Than or Equal to 1:160
Time Frame: 4-Week Dosing Interval (Week 7, Week 19, and Week 31); 3-Week Dosing Interval (Week 4, Week 16, and Week 28)
Population: Epoch 2 Safety Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
percentage of participants | 0

23. Secondary Outcome: Epoch 2: Percentage of Participants Who Develop Neutralizing Antibodies to rHuPH20
Time Frame: 4-Week Dosing Interval (Week 7, Week 19, and Week 31); 3-Week Dosing Interval (Week 4, Week 16, and Week 28)
Population: Epoch 2 Safety Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
percentage of participants | 0

24. Secondary Outcome: Percentage of Participants Who Experienced Tolerability Events Related to the Infusion of TAK-771
Description: Tolerability events is defined as a case that the infusion rate is reduced, or that the infusion is interrupted or stopped, due to a TEAE related to TAK-771 infusion.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16 | 16
percentage of participants | 0 | 0

25. Secondary Outcome: Epoch 1: Number of Weeks to Reach Final Dose Interval (3 Weeks or 4 Weeks)
Description: The number of weeks to reach final dose interval is defined as treatment duration of Epoch 1.
Time Frame: Up to Week 4 for Participants with 4-Week Dosing Interval or Up to Week 3 for Participants with 3-Week Dosing Interval
Population: Safety Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Median (Full Range); unit: weeks
Arm/Group | Epoch 1: TAK-771 Ramp up Period
Number analyzed (Participants) | 16
weeks | 6.00 [3.0 to 6.9]

26. Secondary Outcome: Epoch 2: Percentage of Participants Who Achieve a Treatment Interval of 3 or 4 Weeks
Time Frame: as for outcome 1
Population: Epoch 2 Safety Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
percentage of participants | 100.0

27. Secondary Outcome: Epoch 2: Percentage of Participants Who Maintain a Treatment Interval of 3 or 4 Weeks
Time Frame: as for outcome 1
Population: Epoch 2 Safety Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Number; unit: percenatge of participants
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
percenatge of participants | 100.0

28. Secondary Outcome: Annual Rate of Validated Acute Serious Bacterial Infections (ASBIs) Per Participant Per Year
Description: The annual rate of validated ASBIs is calculated as the mean number of ASBIs per participant per year.
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Mean (Standard Deviation); unit: ASBIs per participant per year
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
ASBIs per participant per year | 0.00 (0.00)

29. Secondary Outcome: Annual Rate of All Infections Per Participant Per Year
Description: The annual rate of all infections is calculated as the mean number of infections per participant per year.
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Mean (Standard Deviation); unit: infections per participant per year
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
infections per participant per year | 2.69 (3.133)

30. Secondary Outcome: Healthcare Resource Utilization: Days Not Able To Attend School/Work or To Perform Normal Daily Activities Due to Illness/Infection
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Median (Full Range); unit: number of days
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
number of days | 0 [0 to 26.8]

31. Secondary Outcome: Healthcare Resource Utilization: Days on Antibiotics
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Median (Full Range); unit: number of days
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
number of days | 0 [0 to 40.2]

32. Secondary Outcome: Healthcare Resource Utilization: Number of Hospitalizations Due to Illness/Infection Per Year
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Mean (Standard Deviation); unit: hospitalizations per year
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
hospitalizations per year | 0.22 (0.591)

33. Secondary Outcome: Healthcare Resource Utilization: Length of Stay in Days of Hospitalizations Due to Illness/Infection Per Participant Per Year
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Median (Full Range); unit: hospitalization days/participant/year
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
hospitalization days/participant/year | 0 [0 to 10.5]

34. Secondary Outcome: Healthcare Resource Utilization: Number of Acute (Urgent or Unscheduled) Physician Visits Due to Illness/Infection
Time Frame: as for outcome 13
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Median (Full Range); unit: Acute Physician Visits
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
Acute Physician Visits | 1.74 [0 to 11.7]

35. Secondary Outcome: Infusion Parameters in Epoch 2: Number of Infusion Sites Per Infusion
Description: Total number of infusion sites injected in Epoch 2 / Total number of infusions administered in Epoch 2.
Time Frame: From Week 7 up to Week 31 for Participants with 4-Week Dosing Interval or From Week 4 up to Week 28 for Participants with 3-Week Dosing Interval
Population: Epoch 2 Full Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Mean (Standard Deviation); unit: infusion sites per infusion
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
infusion sites per infusion | 1.77 (0.394)

36. Secondary Outcome: Infusion Parameters in Epoch 2: Number of Infusion Sites Per Month
Description: Total number of infusion sites injected in Epoch 2 / (duration of Epoch 2 / 30.4375), where duration of Epoch 2 is calculated as the end date of the Epoch 2 - the start date of the Epoch 2 + 1.
Time Frame: as for outcome 35
Population: Epoch 2 Full Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Mean (Standard Deviation); unit: infusion sites per month
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
infusion sites per month | 2.02 (0.514)

37. Secondary Outcome: Infusion Parameters in Epoch 2: Duration of Individual Infusions
Description: End date and time of infusion in Epoch 2 - Start date and time of infusion in Epoch 2, for each infusion per participant.
Time Frame: as for outcome 35
Population: Epoch 2 Full Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Median (Full Range); unit: minutes
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
minutes | 74.0 [18 to 207]

38. Secondary Outcome: Infusion Parameters in Epoch 2: Maximum Infusion Rate Per Site
Description: Maximum Infusion Rate results from CRF / number of infusion sites/body.
Time Frame: as for outcome 35
Population: Epoch 2 Full Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Measure: Mean (Standard Deviation); unit: mL/hour per site
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
mL/hour per site | 222.3 (83.77)

39. Secondary Outcome: Infusion Parameters in Epoch 2: Infusion Volume Per Site
Description: Infusion Volume per Site is scheduled Dose results from CRF / number of infusion sites/body.
Time Frame: as for outcome 35
Population: Epoch 2 Full Analysis Set included all participants who received investigational drug at least once in Epoch 2. Number analyzed are the number of participants with data available for analysis at given timepoint.
Measure: Mean (Standard Deviation); unit: mL/site
Arm/Group | Epoch 2: TAK-771 Full Dose Treatment Period
Number analyzed (Participants) | 16
mL/site | 117.3 (77.73)

40. Secondary Outcome: Quality of Life (QOL): Pediatric Quality of Life Inventory (PEDS-QL)
Description: The PEDS-QL is a generic Health-Related Quality of Life (HR QoL) instrument designed specifically for a pediatric population. It captures the following domains: general health/activities, feelings/emotional, social functioning, school functioning. In this study, 2-7 years (parent as observer), 8-13 years (participant as observer) for PEDS-QL health questionnaire will be analyzed. Higher scores indicate better quality of life (QOL) for all domains of the PEDS-QL. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Four dimensions (physical, emotional, social, & school functioning) are scored.
Time Frame: 4-Week Dosing Interval (Week 1 and Week 31); 3-Week Dosing Interval (Week 1 and Week 28)
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants available for analysis in the specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 5
score on a scale
  Baseline (Week 1), 2-7 years, Total score, 4-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-7 years, Total score, 4-week interval | 93.48 (NA) — Standard deviation is not estimable for single participant
  Baseline (Week 1), 2-7 years, Total score, 3-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-7 years, Total score, 3-week interval | 76.09 (NA) — Standard deviation is not estimable for single participant
  Baseline (Week 1), 8-13 years, Total score, 4-week interval: number analyzed (Participants) | 3
  Baseline (Week 1), 8-13 years, Total score, 4-week interval | 77.17 (18.091)
  Change from Baseline (EOS/ET),2-7 years, Total score, 4-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET),2-7 years, Total score, 4-week interval | 2.17 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET),2-7 years, Total score, 3-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET),2-7 years, Total score, 3-week interval | 11.96 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 8-13 years, Total score, 4-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 8-13 years, Total score, 4-week interval | 11.41 (3.843)

41. Secondary Outcome: QOL: Short Form-36 Health Survey Version 2 (SF-36 v2)
Description: The SF-36 is a generic quality-of-life instrument that has been widely used to assess Health-Related Quality of Life (HR QoL) of participants. In this study, 14 years and older (participant as observer) for SF-36 health questionnaire will be analyzed. Generic instruments are used in general populations to assess a wide range of domains applicable to a variety of health states, conditions, and diseases. The SF-36 consists of 36 items that are aggregated into 8 multi-item scales (physical functioning, role - physical, bodily pain, general health, vitality, social functioning, role - emotional, and mental health), with scores ranging from 0 to 100. Higher scores indicate better HR QoL. Physical component summary (PCS).
Time Frame: 4-Week Dosing Interval (Week 1 and Week 31); 3-Week Dosing Interval (Week 1 and Week 28)
Population: Epoch 2 Full Analysis Set included all participants who received investigational drug at least once in Epoch 2. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants available for analysis in the specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 8
score on a scale
  Baseline (Week 1), 14 years and older, Physical component summary (PCS) score, 4-week interval: number analyzed (Participants) | 6
  Baseline (Week 1), 14 years and older, Physical component summary (PCS) score, 4-week interval | 51.85 (3.458)
  Baseline (Week 1), 14 years and older, Physical component summary (PCS) score, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 14 years and older, Physical component summary (PCS) score, 3-week interval | 53.30 (2.546)
  Baseline (Week 1), 14 years and older, Mental component summary (MCS) score 4-week interval: number analyzed (Participants) | 6
  Baseline (Week 1), 14 years and older, Mental component summary (MCS) score 4-week interval | 51.38 (14.060)
  Baseline (Week 1), 14 years and older, Mental component summary (MCS) score 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 14 years and older, Mental component summary (MCS) score 3-week interval | 59.90 (10.465)
  Baseline (Week 1), >=14 years, Role/social component summary (RCS) score, 4-week interval: number analyzed (Participants) | 6
  Baseline (Week 1), >=14 years, Role/social component summary (RCS) score, 4-week interval | 49.67 (8.495)
  Baseline (Week 1), >=14 years, Role/social component summary (RCS) score, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), >=14 years, Role/social component summary (RCS) score, 3-week interval | 53.50 (8.768)
  Change from Baseline (EOS/ET), >=14 years, Physical component summary (PCS) score, 4-week interval: number analyzed (Participants) | 6
  Change from Baseline (EOS/ET), >=14 years, Physical component summary (PCS) score, 4-week interval | 0.20 (8.709)
  Change from Baseline (EOS/ET), >=14 years, Physical component summary (PCS) score, 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), >=14 years, Physical component summary (PCS) score, 3-week interval | -1.85 (1.202)
  Change from Baseline (EOS/ET), >=14 years, Mental component summary (MCS) score 4-week interval: number analyzed (Participants) | 6
  Change from Baseline (EOS/ET), >=14 years, Mental component summary (MCS) score 4-week interval | -3.12 (5.605)
  Change from Baseline (EOS/ET), >=14 years, Mental component summary (MCS) score 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), >=14 years, Mental component summary (MCS) score 3-week interval | -3.55 (0.636)
  Change from Baseline (EOS/ET), >=14 years, Role/social component summary (RCS) score 4-week interval: number analyzed (Participants) | 6
  Change from Baseline (EOS/ET), >=14 years, Role/social component summary (RCS) score 4-week interval | -0.80 (6.592)
  Change from Baseline (EOS/ET), >=14 years, Role/social component summary (RCS) score,3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), >=14 years, Role/social component summary (RCS) score,3-week interval | 4.90 (3.394)

42. Secondary Outcome: QOL: EuroQoL (Quality of Life)-5 Dimensions 3 Levels (EQ-5D-3L) Health Questionnaire Index Score
Description: The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to all participants to assess the effect of the treatment on the participants' quality of life. Participants select answer for each of the following 3-level dimensions: 1) mobility; 2) self-care; 3) usual activities; 4) pain/discomfort; 5) anxiety/depression used to compute an index score ranging from 0 (worst imaginable health state) to 1 (best imaginable health state). An increase in the EQ-5D-3L index score indicates improvement.
Time Frame: 4-Week dosing interval (Week 1 and Week 31); 3-Week dosing interval (Week 1 and Week 28)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 12
score on a scale
  Baseline (Week 1), 2-11 years, EQ-5D index score, 4-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 2-11 years, EQ-5D index score, 4-week interval | 1.0000 (0.00000)
  Baseline (Week 1), 2-11 years, EQ-5D index score, 3-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-11 years, EQ-5D index score, 3-week interval | 0.6750 (NA) — Standard deviation is not estimable for single participant.
  Baseline (Week 1), 12 years and older, EQ-5D index score, 4-week interval: number analyzed (Participants) | 7
  Baseline (Week 1), 12 years and older, EQ-5D index score, 4-week interval | 0.9271 (0.12655)
  Baseline (Week 1), 12 years and older, EQ-5D index score, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 12 years and older, EQ-5D index score, 3-week interval | 1 (0)
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D index score, 4-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D index score, 4-week interval | 0.0000 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D index score, 3-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D index score, 3-week interval | 0.3250 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D index score, 4-week interval: number analyzed (Participants) | 7
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D index score, 4-week interval | 0.0729 (0.12655)
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D index score, 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D index score, 3-week interval | 0.0000 (0.00000)

43. Secondary Outcome: QOL: EuroQoL (Quality of Life)-5 Dimensions 3 Levels (EQ-5D-3L) Health Questionnaire Visual Analogue Scale (VAS) Score
Description: The EQ-5D-3L is a standardized instrument for use as a measure of health outcome and was administered to all participants to assess the effect of the treatment on the participants' quality of life. The EQ-5D-3L includes a visual analog scale (VAS), a vertical scale that allows the participants to indicate their health state that day, and ranges from 0 (worst imaginable) to 100 (best imaginable), with higher scores indicating better health state.
Time Frame: 4-Week dosing interval (Week 1 and Week 31); 3-Week dosing interval (Week 1 and Week 28)
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 12
score on a scale
  Baseline (Week 1), 2-11 years, EQ-5D VAS score, 4-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 2-11 years, EQ-5D VAS score, 4-week interval | 95.0 (7.07)
  Baseline (Week 1), 2-11 years, EQ-5D VAS score, 3-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-11 years, EQ-5D VAS score, 3-week interval | 100.0 (NA) — Standard deviation is not estimable for single participant.
  Baseline (Week 1), 12 years and older, EQ-5D VAS score, 4-week interval: number analyzed (Participants) | 7
  Baseline (Week 1), 12 years and older, EQ-5D VAS score, 4-week interval | 76.3 (13.24)
  Baseline (Week 1), 12 years and older, EQ-5D VAS score, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 12 years and older, EQ-5D VAS score, 3-week interval | 85.0 (7.07)
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D VAS score, 4-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D VAS score, 4-week interval | -5.0 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D VAS score, 3-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-11 years, EQ-5D VAS score, 3-week interval | -10 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D VAS score, 4-week interval: number analyzed (Participants) | 7
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D VAS score, 4-week interval | 6.3 (9.78)
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D VAS score, 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 12 years and older, EQ-5D VAS score, 3-week interval | -2.5 (3.54)

44. Secondary Outcome: Treatment Preference
Description: Treatment preference questionnaire is a self-administered questionnaire developed to assess participants' preference towards the administration of new subcutaneous immunoglobulin (SCIG) therapy. There are 4-items on the questionnaire, which investigate a participant's preference on the clinic/hospital/home setting of receiving the immunoglobulin (IG) therapy, the participant's rating on the frequency and method of administration, and the participant's preference to continue receiving the IGSC treatment.
Time Frame: as for outcome 1
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 16
Participants
  2-13 years, Before your participation in trial, where did you receive your IG therapy?=At hospital: number analyzed (Participants) | 5
  2-13 years, Before your participation in trial, where did you receive your IG therapy?=At hospital | 4
  2-13 years, Before your participation in the trial, where did you receive your IG therapy?=At home: number analyzed (Participants) | 5
  2-13 years, Before your participation in the trial, where did you receive your IG therapy?=At home | 2
  2-13 years, Where do you prefer to receive your immunoglobulin therapy?=At hospital: number analyzed (Participants) | 5
  2-13 years, Where do you prefer to receive your immunoglobulin therapy?=At hospital | 2
  2-13 years, Where do you prefer to receive your IG therapy?=At home: number analyzed (Participants) | 5
  2-13 years, Where do you prefer to receive your IG therapy?=At home | 1
  2-13 years, Where do you prefer to receive your IG therapy?=No Preference: number analyzed (Participants) | 5
  2-13 years, Where do you prefer to receive your IG therapy?=No Preference | 2
  2-13 years, frequency of administration=Like very much: number analyzed (Participants) | 5
  2-13 years, frequency of administration=Like very much | 3
  2-13 years, frequency of administration=Like: number analyzed (Participants) | 5
  2-13 years, frequency of administration=Like | 1
  2-13 years, Frequency of administration=No Preference: number analyzed (Participants) | 5
  2-13 years, Frequency of administration=No Preference | 1
  2-13 years, number of needlesticks per month=Like very much: number analyzed (Participants) | 5
  2-13 years, number of needlesticks per month=Like very much | 2
  2-13 years, number of needlesticks per month=Like: number analyzed (Participants) | 5
  2-13 years, number of needlesticks per month=Like | 2
  2-13 years, number of needlesticks per month=No preference: number analyzed (Participants) | 5
  2-13 years, number of needlesticks per month=No preference | 1
  2-13 years, total time spent for my treatment per month=Like: number analyzed (Participants) | 5
  2-13 years, total time spent for my treatment per month=Like | 3
  2-13 years, total time spent for my treatment per month=No Preference: number analyzed (Participants) | 5
  2-13 years, total time spent for my treatment per month=No Preference | 2
  2-13 years, ease of administration= Like: number analyzed (Participants) | 5
  2-13 years, ease of administration= Like | 1
  2-13 years, ease of administration= No Preference: number analyzed (Participants) | 5
  2-13 years, ease of administration= No Preference | 3
  2-13 years, The ease of administration= Dislike: number analyzed (Participants) | 5
  2-13 years, The ease of administration= Dislike | 1
  2-13 years, potential to self-administer=Like very much: number analyzed (Participants) | 5
  2-13 years, potential to self-administer=Like very much | 1
  2-13 years, potential to self-administer=No preference: number analyzed (Participants) | 5
  2-13 years, potential to self-administer=No preference | 2
  2-13 years, potential to self-administer=Dislike: number analyzed (Participants) | 5
  2-13 years, potential to self-administer=Dislike | 1
  2-13 years, potential to self-administer=Dislike very much: number analyzed (Participants) | 5
  2-13 years, potential to self-administer=Dislike very much | 1
  2-13 years, ability to fit my treatment into my own schedule= Like: number analyzed (Participants) | 5
  2-13 years, ability to fit my treatment into my own schedule= Like | 3
  2-13 years, ability to fit my treatment into my own schedule= No Preference: number analyzed (Participants) | 5
  2-13 years, ability to fit my treatment into my own schedule= No Preference | 2
  2-13 years, overall convenience=Like: number analyzed (Participants) | 5
  2-13 years, overall convenience=Like | 4
  2-13 years, overall convenience=No preference: number analyzed (Participants) | 5
  2-13 years, overall convenience=No preference | 1
  2-13 years, amount of time administration takes=Like: number analyzed (Participants) | 5
  2-13 years, amount of time administration takes=Like | 2
  2-13 years, amount of time administration takes=No preference: number analyzed (Participants) | 5
  2-13 years, amount of time administration takes=No preference | 2
  2-13 years, amount of time administration takes=Dislike: number analyzed (Participants) | 5
  2-13 years, amount of time administration takes=Dislike | 1
  2-13 years, complexity of administration process=Like: number analyzed (Participants) | 5
  2-13 years, complexity of administration process=Like | 2
  2-13 years, complexity of administration process=No preference: number analyzed (Participants) | 5
  2-13 years, complexity of administration process=No preference | 2
  2-13 years, complexity of administration process=Dislike: number analyzed (Participants) | 5
  2-13 years, complexity of administration process=Dislike | 1
  2-13 years, My ability to self-administer without medical supervision=Like very much: number analyzed (Participants) | 5
  2-13 years, My ability to self-administer without medical supervision=Like very much | 1
  2-13 years, My ability to self-administer without medical supervision=No preference: number analyzed (Participants) | 5
  2-13 years, My ability to self-administer without medical supervision=No preference | 1
  2-13 years, My ability to self-administer without medical supervision=Dislike: number analyzed (Participants) | 5
  2-13 years, My ability to self-administer without medical supervision=Dislike | 1
  2-13 years, My ability to self-administer without medical supervision=Dislike very much: number analyzed (Participants) | 5
  2-13 years, My ability to self-administer without medical supervision=Dislike very much | 2
  2-13 years, would you choose to continue receiving your treatment using IGg10% with rHuPH20 SC?=Yes: number analyzed (Participants) | 5
  2-13 years, would you choose to continue receiving your treatment using IGg10% with rHuPH20 SC?=Yes | 5
  14 years and older, Before your participation, where did you receive your IG therapy?=At hospital: number analyzed (Participants) | 11
  14 years and older, Before your participation, where did you receive your IG therapy?=At hospital | 8
  14 years and older, Before your participation, where did you receive your IG therapy?=At home: number analyzed (Participants) | 11
  14 years and older, Before your participation, where did you receive your IG therapy?=At home | 7
  14 years and older, Before your participation, where did you receive your IG therapy?=Other: number analyzed (Participants) | 11
  14 years and older, Before your participation, where did you receive your IG therapy?=Other | 1
  14 years and older, Where do you prefer to receive your IG therapy? = At hospital: number analyzed (Participants) | 11
  14 years and older, Where do you prefer to receive your IG therapy? = At hospital | 2
  14 years and older, Where do you prefer to receive your IG therapy? = At home: number analyzed (Participants) | 11
  14 years and older, Where do you prefer to receive your IG therapy? = At home | 7
  14 years and older, Where do you prefer to receive your IG therapy? = No preference: number analyzed (Participants) | 11
  14 years and older, Where do you prefer to receive your IG therapy? = No preference | 2
  14 years and older, frequency of administration=Like very much: number analyzed (Participants) | 11
  14 years and older, frequency of administration=Like very much | 3
  14 years and older, frequency of administration=Like: number analyzed (Participants) | 11
  14 years and older, frequency of administration=Like | 7
  14 years and older, frequency of administration=No preference: number analyzed (Participants) | 11
  14 years and older, frequency of administration=No preference | 1
  14 years and older, number of needlesticks per month=Like: number analyzed (Participants) | 11
  14 years and older, number of needlesticks per month=Like | 8
  14 years and older, number of needlesticks per month=No preference: number analyzed (Participants) | 11
  14 years and older, number of needlesticks per month=No preference | 3
  14 years and older, total time spent for my treatment per month = Like very much: number analyzed (Participants) | 11
  14 years and older, total time spent for my treatment per month = Like very much | 1
  14 years and older, total time spent for my treatment per month=Like: number analyzed (Participants) | 11
  14 years and older, total time spent for my treatment per month=Like | 6
  14 years and older, total time spent for my treatment per month=No preference: number analyzed (Participants) | 11
  14 years and older, total time spent for my treatment per month=No preference | 2
  14 years and older, total time spent for my treatment per month=Dislike: number analyzed (Participants) | 11
  14 years and older, total time spent for my treatment per month=Dislike | 2
  14 years and older, ease of administration=Like: number analyzed (Participants) | 11
  14 years and older, ease of administration=Like | 2
  14 years and older, ease of administration=No preference: number analyzed (Participants) | 11
  14 years and older, ease of administration=No preference | 2
  14 years and older, ease of administration=Dislike: number analyzed (Participants) | 11
  14 years and older, ease of administration=Dislike | 6
  14 years and older, ease of administration=Dislike very much: number analyzed (Participants) | 11
  14 years and older, ease of administration=Dislike very much | 1
  14 years and older, potential to self-administer=Like: number analyzed (Participants) | 11
  14 years and older, potential to self-administer=Like | 8
  14 years and older, The potential to self-administer = No preference: number analyzed (Participants) | 11
  14 years and older, The potential to self-administer = No preference | 1
  14 years and older, potential to self-administer=Dislike: number analyzed (Participants) | 11
  14 years and older, potential to self-administer=Dislike | 1
  14 years and older, potential to self-administer=Dislike very much: number analyzed (Participants) | 11
  14 years and older, potential to self-administer=Dislike very much | 1
  14 years and older, ability to fit my treatment into my own schedule= Like very much: number analyzed (Participants) | 11
  14 years and older, ability to fit my treatment into my own schedule= Like very much | 1
  14 years and older, ability to fit my treatment into my own schedule= Like: number analyzed (Participants) | 11
  14 years and older, ability to fit my treatment into my own schedule= Like | 7
  14 years and older, ability to fit my treatment into my own schedule= No preference: number analyzed (Participants) | 11
  14 years and older, ability to fit my treatment into my own schedule= No preference | 2
  14 years and older, ability to fit my treatment into my own schedule= Dislike: number analyzed (Participants) | 11
  14 years and older, ability to fit my treatment into my own schedule= Dislike | 1
  14 years and older, overall convenience = Like: number analyzed (Participants) | 11
  14 years and older, overall convenience = Like | 8
  14 years and older, overall convenience = No preference: number analyzed (Participants) | 11
  14 years and older, overall convenience = No preference | 2
  14 years and older, overall convenience = Dislike: number analyzed (Participants) | 11
  14 years and older, overall convenience = Dislike | 1
  14 years and older, amount of time administration takes = Like: number analyzed (Participants) | 11
  14 years and older, amount of time administration takes = Like | 7
  14 years and older, amount of time administration takes = No preference: number analyzed (Participants) | 11
  14 years and older, amount of time administration takes = No preference | 3
  14 years and older, amount of time administration takes = Dislike: number analyzed (Participants) | 11
  14 years and older, amount of time administration takes = Dislike | 1
  14 years and older, complexity of administration process=Like very much: number analyzed (Participants) | 11
  14 years and older, complexity of administration process=Like very much | 1
  14 years and older, complexity of administration process=Like: number analyzed (Participants) | 11
  14 years and older, complexity of administration process=Like | 1
  14 years and older, complexity of administration process=No preference: number analyzed (Participants) | 11
  14 years and older, complexity of administration process=No preference | 2
  14 years and older, complexity of administration process=Dislike: number analyzed (Participants) | 11
  14 years and older, complexity of administration process=Dislike | 6
  14 years and older, complexity of administration process=Dislike very much: number analyzed (Participants) | 11
  14 years and older, complexity of administration process=Dislike very much | 1
  14 years and older, My ability to self-administer without medical supervision=Like very much: number analyzed (Participants) | 11
  14 years and older, My ability to self-administer without medical supervision=Like very much | 1
  14 years and older, My ability to self-administer without medical supervision=Like: number analyzed (Participants) | 11
  14 years and older, My ability to self-administer without medical supervision=Like | 6
  14 years and older, My ability to self-administer without medical supervision = No preference: number analyzed (Participants) | 11
  14 years and older, My ability to self-administer without medical supervision = No preference | 1
  14 years and older, My ability to self-administer without medical supervision = Dislike: number analyzed (Participants) | 11
  14 years and older, My ability to self-administer without medical supervision = Dislike | 2
  14 years and older, My ability to self-administer without medical supervision = Dislike very much: number analyzed (Participants) | 11
  14 years and older, My ability to self-administer without medical supervision = Dislike very much | 1
  14 years and older, choose to continue receiving your treatment using IGg 10% with rHuPH20 SC?=Yes: number analyzed (Participants) | 11
  14 years and older, choose to continue receiving your treatment using IGg 10% with rHuPH20 SC?=Yes | 9
  14 years and older, choose to continue receiving your treatment using IGg 10% with rHuPH20 SC?= No: number analyzed (Participants) | 11
  14 years and older, choose to continue receiving your treatment using IGg 10% with rHuPH20 SC?= No | 2

45. Secondary Outcome: Treatment Satisfaction: Questionnaire for Medication-9 (TSQM-9)
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. In this study, 2-12 years (parent as observer), 13 years and older (participant as observer) for TSQM health questionnaire will be analyzed. TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain.
Time Frame: 4-Week dosing interval (Week 1 and Week 31); 3-Week dosing interval (Week 1 and Week 28)
Population: Full Analysis Set included all enrolled participants who received investigational drug at least once. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 and 2
Number analyzed (Participants) | 12
score on a scale
  Baseline (Week 1), 2-12 years, Effectiveness, 4-week interval: number analyzed (Participants) | 3
  Baseline (Week 1), 2-12 years, Effectiveness, 4-week interval | 64.81 (3.208)
  Baseline (Week 1), 2-12 years, Effectiveness, 3-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-12 years, Effectiveness, 3-week interval | 94.44 (NA) — Standard deviation is not estimable for single participant.
  Baseline (Week 1), 2-12 years, Convenience, 4-week interval: number analyzed (Participants) | 3
  Baseline (Week 1), 2-12 years, Convenience, 4-week interval | 44.44 (19.245)
  Baseline (Week 1), 2-12 years, Convenience, 3-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-12 years, Convenience, 3-week interval | 38.89 (NA) — Standard deviation is not estimable for single participant.
  Baseline (Week 1), 2-12 years, Global satisfaction, 4-week interval: number analyzed (Participants) | 3
  Baseline (Week 1), 2-12 years, Global satisfaction, 4-week interval | 59.52 (10.911)
  Baseline (Week 1), 2-12 years, Global satisfaction, 3-week interval: number analyzed (Participants) | 1
  Baseline (Week 1), 2-12 years, Global satisfaction, 3-week interval | 100.00 (NA) — Standard deviation is not estimable for single participant.
  Baseline (Week 1), 13 years and older, Effectiveness, 4-week interval: number analyzed (Participants) | 6
  Baseline (Week 1), 13 years and older, Effectiveness, 4-week interval | 64.81 (18.812)
  Baseline (Week 1), 13 years and older, Effectiveness, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 13 years and older, Effectiveness, 3-week interval | 63.89 (3.928)
  Baseline (Week 1), 13 years and older, Convenience, 4-week interval: number analyzed (Participants) | 6
  Baseline (Week 1), 13 years and older, Convenience, 4-week interval | 62.04 (19.694)
  Baseline (Week 1), 13 years and older, Convenience, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 13 years and older, Convenience, 3-week interval | 44.44 (0.000)
  Baseline (Week 1), 13 years and older, Global satisfaction, 4-week interval: number analyzed (Participants) | 6
  Baseline (Week 1), 13 years and older, Global satisfaction, 4-week interval | 60.71 (8.748)
  Baseline (Week 1), 13 years and older, Global satisfaction, 3-week interval: number analyzed (Participants) | 2
  Baseline (Week 1), 13 years and older, Global satisfaction, 3-week interval | 64.29 (10.102)
  Change from Baseline (EOS/ET), 2-12 years, Effectiveness, 4-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 2-12 years, Effectiveness, 4-week interval | 0.00 (0.000)
  Change from Baseline (EOS/ET), 2-12 years, Effectiveness, 3-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-12 years, Effectiveness, 3-week interval | -27.78 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 2-12 years, Convenience, 4-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 2-12 years, Convenience, 4-week interval | 13.89 (3.928)
  Change from Baseline (EOS/ET), 2-12 years, Convenience, 3-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-12 years, Convenience, 3-week interval | 0.00 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 2-12 years, Global satisfaction, 4-week interval: number analyzed (Participants) | 3
  Change from Baseline (EOS/ET), 2-12 years, Global satisfaction, 4-week interval | 10.71 (5.051)
  Change from Baseline (EOS/ET), 2-12 years, Global satisfaction, 3-week interval: number analyzed (Participants) | 1
  Change from Baseline (EOS/ET), 2-12 years, Global satisfaction, 3-week interval | -28.57 (NA) — Standard deviation is not estimable for single participant.
  Change from Baseline (EOS/ET), 13 years and older, Effectiveness, 4-week interval: number analyzed (Participants) | 6
  Change from Baseline (EOS/ET), 13 years and older, Effectiveness, 4-week interval | -12.04 (26.156)
  Change from Baseline (EOS/ET), 13 years and older, Effectiveness, 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 13 years and older, Effectiveness, 3-week interval | 2.78 (3.928)
  Change from Baseline (EOS/ET), 13 years and older, Convenience, 4-week interval: number analyzed (Participants) | 6
  Change from Baseline (EOS/ET), 13 years and older, Convenience, 4-week interval | -3.70 (20.688)
  Change from Baseline (EOS/ET), 13 years and older, Convenience, 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 13 years and older, Convenience, 3-week interval | 0.00 (7.857)
  Change from Baseline (EOS/ET), 13 years and older, Global satisfaction, 4-week interval: number analyzed (Participants) | 6
  Change from Baseline (EOS/ET), 13 years and older, Global satisfaction, 4-week interval | -13.10 (26.885)
  Change from Baseline (EOS/ET), 13 years and older, Global satisfaction, 3-week interval: number analyzed (Participants) | 2
  Change from Baseline (EOS/ET), 13 years and older, Global satisfaction, 3-week interval | -3.57 (5.051)

ADVERSE EVENTS:
Time Frame: From study start up to Week 28 for the 3-week dosing intervals and up to Week 31 for 4-week dosing intervals
Description: Safety analysis set included all enrolled participants who received investigational drug at least once. Epoch 2 Safety Analysis Set included all participants who received investigational drug at least once in Epoch 2.
Groups:
- Epoch 2: TAK-771 Full Dose Treatment Period: TAK-771 included IGI 10% and rHuPH20. Participants received subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3, or 4 weeks for up to Week 24.
Arm/Group | Epoch 1: TAK-771 Ramp up Period | Epoch 2: TAK-771 Full Dose Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/16
Other Adverse Events (participants affected / at risk) | 13/16 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1: TAK-771 Ramp up Period (N=16) | Epoch 2: TAK-771 Full Dose Treatment Period (N=16)
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1: TAK-771 Ramp up Period (N=16) | Epoch 2: TAK-771 Full Dose Treatment Period (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Administration site pain (General disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Application site erythema (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2
Chronic sinusitis (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Infusion site erythema (General disorders) | 2 | 2
Infusion site pain (General disorders) | 2 | 0
Infusion site swelling (General disorders) | 2 | 1
Injection site erythema (General disorders) | 2 | 2
Injection site induration (General disorders) | 0 | 1
Injection site pain (General disorders) | 2 | 2
Injection site pruritus (General disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Malaise (General disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3
Ocular hyperaemia (Eye disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Peripheral swelling (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Vaccination site pain (General disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05150340/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT05150340/SAP_001.pdf